CLINICAL TRIAL: NCT02858583
Title: SURV1VE-Trial - Sustained Inflation and Chest Compression Versus 3:1 Chest Compression to Ventilation Ratio During Cardiopulmonary Resuscitation of Asphyxiated Newborns: A Randomized Controlled Trial
Brief Title: SI + CC Versus 3:1 C:V Ratio During Neonatal CPR
Acronym: SURV1VE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.0
Record Dates: First submitted 2016-07-30; First posted 2016-08-08 (Estimated); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Heart Arrest; Birth Asphyxia; Bradycardia
Keywords: Chest Compression; Newborn; Infant; Sustained Inflation
MeSH Terms: conditions — Heart Arrest; Asphyxia Neonatorum; Bradycardia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (CC+SI) (Experimental): Infants randomized into the "CC+SI group" will receive a SI with a PIP of 25-30 cmH2O while receiving chest compression. The SI will be delivered over a period of 45 seconds. This will be followed by PEEP of 5-8 cm water to perform an assessment of the newborn's heart rate. If heart rate is >60/min continue with standard care as per local hospital policy (standard hospital practice guideline). If heart rate remains <60/min continue with CC+SI for another 45sec at which time a further assessment should be performed. If heart rate remains <60/min continue with CC+SI.
  Interventions: Procedure: CC+SI
- Control (3:1 C:V) (Active Comparator): Infants randomized into the "3:1 C:V group" will receive CC at a rate of 90/min and 30 ventilations/min in a 3:1 C:V ratio as recommended by the current resuscitation guidelines.
  Interventions: Procedure: 3:1 C:V

INTERVENTIONS:
Procedure: CC+SI — chest compression will be delivered during sustained inflation (CC+SI). The duration of each sustain inflation is 20sec. After 20sec a pause of 1sec id done before the next sustained inflation is delivered for another 20sec. Chest compressions are given continuously. This approach is continued until return of spontaneous circulation.
  Arms: Intervention (CC+SI)
Procedure: 3:1 C:V — During 3:1 C:V. 3 chest compressions are given, then stopped and then 1 inflation is given. This approach is continued until return of spontaneous circulation.
  Arms: Control (3:1 C:V)

SUMMARY:
Research question In newborn infants requiring CPR, does CC superimposed by sustained inflation compared to 3:1 compression to ventilation ratio improves return of spontaneous circulation?

Overall objective: CC superimposed by sustained inflation will improve short- and long-term outcomes in preterm (>28 weeks or older) and term newborns.

Hypothesis to be tested Primary hypothesis: By using CC superimposed by sustained inflation (CC+SI) during CPR the time needed to achieve return of spontaneous circulation (ROSC) compared to the current 3:1 compression to ventilation (C:V) will be reduced in asphyxiated newborns.

DETAILED DESCRIPTION:
Background The majority of newborn infants successfully make the transition from fetal to neonatal life without any help. However, an estimated 10% of newborns need help to establish effective ventilation, which remains the most critical step of neonatal resuscitation. Fortunately, the need for chest compression (CC) or medications in the delivery room (DR) is rare. Although, only about 0.1% of term infants and up to 15% of preterm infants receive these interventions, this will result in approximately 1 million newborn deaths annually worldwide. A recent cohort study at a level III center with a trained resuscitation team showed that only 6 per 10,000 infants received epinephrine. However, the same study showed that those infants who received epinephrine during resuscitation had a high incidence of mortality (41%) and short-term neurologic morbidity (57% hypoxic-ischemic encephalopathy and seizures)4. A recent review of newborns who received prolonged CC and epinephrine but had no signs of life at 10 minutes following birth noted 83% mortality, with 93% of survivors suffering moderate-to-severe disability. The poor prognosis associated with receiving CC alone or with medications in the DR raises questions as to whether improved cardiopulmonary resuscitation (CPR) methods specifically tailored to the newborn could improve outcomes.

The inability to predict which newborns need CPR, and the infrequent use of CPR in the DR have limited neonatologists' ability to perform rigorous clinical studies to determine the best method for delivering CC to newborn infants. The main cause of cardiovascular collapse in most newborns is asphyxia, which makes newborn infants distinctively different to the adult population. The International Liaison Committee on Resuscitation and the American Academy of Pediatrics/American Heart Association Neonatal Resuscitation Program have recognize this difference, however the guidelines almost exclusively rely on data from studies in the adult population or animal studies. Such data may not be wholly applicable to the neonatal population because the most common cause of cardiovascular collapse in the adult is ventricular fibrillation, not asphyxia. Thus, further studies are needed to determine the optimal method for improving hemodynamics and recovery during neonatal resuscitation.

Research question In newborn infants (preterm infants >28 weeks' gestation and term infants) requiring CPR, does CC during sustained inflation compared to 3:1 compression to ventilation ratio improves return of spontaneous circulation (ROSC)?

Primary objective: To prove that CC during sustained inflation will improve recovery from CPR in preterm and term newborns with faster ROSC than that by 3:1 CPR technique.

Secondary objectives: To examine i) if CC during sustained inflation will improve short- and long-term outcomes in preterm and term newborns, and ii) the value of feedback devices (e.g. ECO2, ECG and/or SpO2) in determining ROSC.

Hypotheses to be tested Primary hypothesis: By using CC during sustained inflation (CC+SI) during CPR the time needed to achieve ROSC compared to the current 3:1 compression to ventilation (C:V) ratio will be reduced in asphyxiated newborns.

Secondary hypotheses: The benefits associated with CC+SI will i) decrease death; ii) improve short- and long-term outcomes in preterm and term newborns; and iii) feedback devices help to determine ROSC.

Methodology Ethics This multi-center cluster randomized clinical trial will be reviewed by the appropriate Research Ethics Office at all participating sites. We will request a deferred consent model at all sites (see parental consent paragraph for details). Written consent will be sought from the parents of these infants as soon as possible after the birth so that acquired data could be utilized for research35.

Inclusion criteria All infants (term or preterm infants >28 weeks' gestation) requiring CC in the delivery room will be eligible for the trial.

Exclusion criteria Infants will be excluded if they have a congenital abnormality or condition that might have an adverse effect on breathing or ventilation (e.g. congenital diaphragmatic hernia), or congenital heart disease requiring intervention in the neonatal period. Infants will be also excluded if their parents refuse to give consent to this study.

Randomization At the beginning of the trial participating sites will be randomized. Centers will be equally allocated to either CC+SI group ("intervention group") or 3:1 C:V group ("control group") for the first year. For the second year, after a wash out period of 2 months, centers in the intervention group will be changed to control and vice versa.

Sample Size and Power calculation Our primary outcome measure will be time to achieve ROSC. We hypothesize that the time to achieve ROSC will be reduced in the "CC+SI group". A sample size of 208 infants, 104 in each group, would be sufficient to detect a clinically important 33% reduction in time to achieve ROSC using Cox proportional hazards regression with 80% power and a 2-tailed alpha error of 0.05. This 33% reduction represents 282 sec versus 420 sec of CC (based on the database of 30 term infants requiring CC in 2014 and 2015 at the Royal Alexandra Hospital, Edmonton). To account for cluster randomization, the sample size is multiplied by design effect of 1.045, so the total sample size is 218 infants, 109 in each group.

Blinding There will be no blinding during the recruitment phase. Each hospital is allocated to one treatment arm and therefore the CC technique used at each particular site is known to the clinical team. The outcome assessor will be unaware of the group allocation. This blinding will be maintained until the data is locked for the final analysis and un-blinded.

Technique of Resuscitation Infants will only be eligible and randomized if they require chest compressions. The methods described below also describe resuscitation interventions for infants prior to the start of chest compressions.

Description of general interventions Term infants The initial steps of the resuscitation will be according to the current neonatal resuscitation guidelines1. Delayed cord clamping should be performed as per local hospital policy (standard hospital practice guideline) at participating sites where eligible. Afterwards, dry and stimulate the infant, and open the airway. If heart rate is <100/min, the infant is gasping or has apnea, start positive pressure ventilation. At the same time consider attaching a pulse oximeter and also consider applying electrocardiography. If heart rate remains <100/min, perform MR. SOPA (Mask is tightly applied to the face, Re-position the head into the "sniffing" orientation, Suction the nares and the pharynx, Open the mouth, Pressure of PPV can be increased to a max of 40 cm H2O, Alternate airway (endotracheal tube or Laryngeal Mask Airway). If heart rate is <60/min or remains <60 despite all steps of MR. SOPA including alternate airway, start chest compressions and increase to 100% oxygen.

Preterm infants The initial steps of the resuscitation will be according to the current neonatal resuscitation guidelines1. Delayed cord clamping should be performed as per local hospital policy (standard hospital practice guideline) at participating sites where eligible. Immediately afterwards, preterm infants (according to local hospital policy - standard hospital practice guideline) will be either placed (without drying) in a polyethylene bag under radiant heat44 or dried and placed under radiant heat.

A pulse oximeter will be used to monitor oxygen saturation immediately after birth and oxygen delivery will be guided by published norm values for oxygen saturation in preterm infants45.

If heart rate is <100/min, the infant is gasping or has apnea, start positive pressure ventilation. Also consider applying electrocardiography at that time. If heart rate remains <100/min, perform MR. SOPA (Mask is tightly applied to the face, Re-position the head into the "sniffing" orientation, Suction the nares and the pharynx, Open the mouth, Pressure of PPV can be increased to a max of 40 cm H2O, Alternate airway (endotracheal tube or Laryngeal Mask Airway). If heart rate is <60/min or remains <60 despite all steps of MR. SOPA start chest compression and increase to 100% oxygen.

Mask Ventilation The clinical team will determine if an infant requires mask ventilation. If mask ventilation is required, it should be provided with a T-Piece device (e.g. Fisher & Paykel, Auckland, New Zealand or Giraffe Warmer, GE Health Care, Burnaby, BC, Canada), and appropriate face mask with default settings for peak inflation pressure (PIP) of 25 cmH2O, a peep expiratory pressure (PEEP) of 5 cm H2O, and a gas flow rate of 8-10L/min using a ventilation rate of 40-60 inflations/min. Initial respiratory support can include initial sustained inflations (instead of positive pressure ventilation alone) as per local hospital policy (standard hospital practice guideline).

Cardiopulmonary Resuscitation If heart rate is <60/min or remains <60/min despite all steps of MR. SOPA start chest compressions. Prior to the start of CC intubation should be considered. However, in cases of intubation failure it is possible to start CC during mask ventilation. Compressions will be performed using the 2-thumb encircling technique as recommended by current resuscitation guidelines46. Epinephrine will be administered according to current resuscitation guidelines either via umbilical vein catheter (0.01 mg/kg per dose - first line) or via endotracheal tube (0.05 mg/kg to 0.1 mg/kg) or every three to five minutes as needed44. Chest compressions and epinephrine will be continued until ROSC.

Determination of ROSC ROSC will defined as an increase in heart rate >60/min for 60sec determined by auscultation of the heart. Return of spontaneous circulation will be assessed after 60sec of a heart rate of >60/min.

The current neonatal resuscitation guidelines do not recommend feedback devices (e.g. exhaled carbon dioxide (ECO2) monitors, electrocardiography (ECG), or pulse oximetry for detection of ROSC1. A secondary objective of the study will be to examine if either feedback device ECO2, ECG or pulse oximetry can be used for detection of ROSC. Participating centres (e.g. Edmonton, Graz, Winnipeg, Ulm, San Diego) are using either ECO2 monitors, ECG, and/or pulse oximetry routinely during neonatal resuscitation35,47-49.

Interventions "3:1 C:V group" If the PIP has been increased >30 cm H2O during MR.SOPA, the PIP should be decreased to 30 cmH2O prior start of chest compression. Infants randomized into the "3:1 C:V group" will receive CC at a rate of 90/min and ventilations at a rate of 30 /min in a 3:1 C:V ratio as recommended by the current resuscitation guidelines1 (study flow diagram). During CC, the inflations should be delivered using a PIP of 25-30 cmH2O (As per local hospital policy /standard hospital practice guideline). Heart rate should be reevaluated every 60sec according to current neonatal resuscitation guidelines1.

"CC+SI group" If the PIP has been increased >30 cm H2O during MR.SOPA, the PIP should be decreased to 30 cmH2O prior start of chest compression. Infants randomized into the "CC+SI group" will receive a SI with a PIP 25-30 cmH2O while receiving CC. CC will be performed at a rate of 90/min. The SI will be delivered over a period of 20 seconds. This will be followed by PEEP of 5-8 cm water as per local hospital policy (standard hospital practice guideline) for one second. Then the next SI for 20sec is started while CCs are continued. Again after 20sec there will be a 1sec pause with PEEP, which will be followed by another SI for 20sec with continuous CC. After 3x20sec SI+CC (total of 60sec) an assessment of heart rate should be performed. If heart rate is >60/min continue with standard care as per local hospital policy (standard hospital practice guideline). If heart rate remains <60/min continue with CC+SI for another 60sec (3x20sec SI+CC (total of 60sec) at which time a further assessment should be performed. If heart rate remains <60/min continue with CC+SI. If CPR is ongoing for 5 minutes using SI+CC, the clinical team must convert to the standard method of care using 3:1 C:V ratio.

Discontinuing Resuscitation Deciding how long resuscitative efforts should continue in any of the study infants will be solely at the discretion of the clinical team in accordance with the current neonatal resuscitation guidelines1 and per local hospital policy (standard hospital practice guideline) at every participating site.

18-24 months follow-up SI+CC might result in improved pCO2 during CPR. A more favourable pCO2 might be neuro-protective, and we hypothesize that SI+CC infants will have a better neurodevelopmental outcome compared to infants randomized to 3:1 C:V. Most infants who receive chest compressions are routinely assessed for neurodevelopmental outcomes at 18-24 months of age in the outpatient clinic in the study hospital. A Bayley III assessment (reference) will be performed by a psychologist or other professional with the relevant competence at the study site. This participant data will be collected at the 18-24 month follow up visit if this is part of routine care; it is not mandatory to collect.

Outcome measures Primary outcome Time to achieve ROSC is defined as a heart rate of >60/min for 60sec determined by auscultation of the heart. Return of spontaneous circulation will be assessed after 60sec of a heart rate of >60/min.

Secondary outcomes Secondary outcomes amongst others will include neonatal mortality (Neonatal death <28 days) and morbidities, for example, rates of brain injury (reported either via magnetic resonance imaging (MRI) or head ultrasound), changes in regional cerebral oxygen saturation using near-infrared spectroscopy (NIRS) monitoring started in the DR and discontinued when clinical stabilization is achieved, results of amplitude-integrated electroencephalograpy (aEEG) monitoring until normalization of background patterns and occurrence of sleep-wake cycling, DR interventions (including the use of epinephrine), admission temperature, use of therapeutic cooling, mechanical ventilation, pneumothorax, use of inotropes, infection/sepsis, intraventricular hemorrhages, necrotizing enterocolitis, bronchopulmonary dysplasia, retinopathy of prematurity and long-term neurodevelopmental outcomes. We will also assess the value of ECO2, ECG and/or SpO2 in determining ROSC as described previously.

Outcome assessment tools Mortality: All causes of mortality will be recorded. Cerebral injury will be assessed with either cerebral ultrasound or cerebral MRI if performed prior to discharge. If an infant dies prior to any neuro-imaging, a request for autopsy should be made. Autopsy could include imaging alone or full autopsy. Morbidity: Case history until discharge or term age (for preterm infants). Secondary outcome parameters: Case history and output from feedback devices.

Compliance with the Protocol The clinical investigation will be conducted in compliance with this protocol. Modifications to the protocol will not be implemented without agreement from the Principal Investigators and relevant ethics committee approval are obtained.

Investigators are not allowed to deviate from the protocol except as specified above. Any major or safety related deviations will be recorded, analyzed and the ethics committees notified. If an investigator refuses to comply with the protocol he/she will be disqualified.

Data collection Infants will be recruited over a period of 26 months. Approximately another six months will be required to collect hospital data on all infants enrolled. Resuscitation data will be collected on a standard form (Neonatal Resuscitation Record) that will form part of each infant's hospital record. The Neonatal Resuscitation Record should be completed by the clinical team attending the resuscitation. Other medical data on each infant will be collected on an electronic Case Report Form (eCRF). The eCRF will be designed in collaboration with Women and Children's Health Research Institute, University of Alberta, Edmonton, Canada. Data will be entered into REDCap database from each site within one week after discharge or death of an infant. Long-term follow-up will be entered within two weeks after examination. All information entered into REDCap database will be used for analysis.

Data analysis The Clinical Research Informatics Core and Biostatistics Core of the Women and Children's Health Research Institute, at the University of Alberta, will do data management and analysis. Additional information about the storage, management and analysis of study data is available.

All analyses will be carried out according to the intention-to-treat principle. Statistical analyses will be performed using IBM SPSS Statistics Ver. 24 (IBM Corp.) and SAS version 9.4 (SAS Institute Inc.) or later.

Interim Analysis Interim safety analysis will be performed at 10%, 25% and 50% of enrolment to review the primary outcome, ROSC, and severe adverse events (SAEs).

Thus, three interim analyses will be performed at 22 patients (11 patients per group), 54 (27 patients per group), and 110 (55 patients per group) to evaluate the efficacy of the intervention. At each interim analysis posterior probability of SI+CC arm to reduce time to ROSC by 10% or more compared to the control arm will be calculated. If this probability is less than 0.5, the trial will be stopped for futility. If the posterior probability is greater than 0.98, the Data and Safety Monitoring Board will consider the trial to be stopped for superiority. Since no statistical tests will be performed at interim analyses, type I error (alpha) does not need adjustment.

Final Analysis Primary Analysis The primary outcome is the time to achieve ROSC defined as a heart rate of >60/min for 60sec. Data will be analyzed on an intention-to treat basis and will include all randomized participants. A per protocol analysis will also be conducted using the data from the actual allocation of participating infants. A survival analysis will be used to analyze the difference in time to ROSC between intervention and control groups. To account for cluster randomization, Cox proportional hazards regression with time to ROSC as an outcome and allocation group as an independent variable will be created. Centers will be entered as clusters in the model and the statistical significance of the allocation group variable will be evaluated. The analysis will be 2-sided and p-value < 0.05 will be considered statistically significant.

Secondary Analysis The data will be presented as mean (standard deviation, SD) for normally distributed continuous variables and median (interquartile range, IQR) when the distribution is skewed. The clinical characteristics and outcome parameters will be compared using Student's t-test for parametric and Mann-Whitney U-test for nonparametric comparisons of continuous variables, and χ2 for categorical variables. All p-values will be 2-sided and p <0.05 will be considered statistically significant.

Assessment of safety Adverse and Serious Adverse Events Infants who require CPR in the DR are a very seriously ill patient group. Most adverse events may be of a serious nature with or without the SURV1VE-trial intervention, and both intervention groups are expected to have a very high proportion of serious adverse events (SAEs). Serious adverse events to be recorded are therefore mortality within the DR (e.g. did not achieve ROSC or did achieve ROSC but care was withdrawn), and within the NICU (any mortality).

Expected adverse events Adverse events we expect to be related to the application of the treatment guideline include: No ROSC leading to death, accidental displacement of the endotracheal tube or extubation, accidental displacement of venous or arterial catheters, use of Nitric Oxide for pulmonary hypertension, sepsis, pneumothorax, and intraventricular hemorrhage (grades 1-4)52.

Data and Safety Monitoring Board A Data and Safety Monitoring Board (DSMB) will monitor the study to: (1) protect all study patients, (2) safeguard the interests of all study patients, (3) monitor the overall conduct of the trial, (4) advise the investigators in order to protect the integrity of the trial, and (5) supervise the conduct and analysis of all interim analyses. To its end the DSMB will receive regular reports from the trial on any injuries or adverse events, any developments that jeopardize the continued success of the trial, and data by which to accomplish the evaluation of pre-determined early stopping rules. Serious Adverse Events to be reported (mortality) will be sent within 72 hours to the DSMB; reports of other/less serious adverse events and recruitment will be sent monthly; demographics and adverse events (including pneumothorax, and intraventricular hemorrhage grade 3 or higher according to Papile52) will be included with the interim and final safety and efficacy analyses. The DSMB will perform interim safety analysis at 10%, 25% and 50% of enrolment to review the primary outcome of ROSC, and SAEs. At the discretion of the DSMB further interim analyses can be requested.

Members of the DSMB are Myra Wyckoff (current Chair of the International Liaison Committee on Resuscitation (ILCOR), Neil Finer (Professor Emeritus, University of California San Diego), and Maryna Yaskina (Statistician, Biostatistics Unit, Women and Children's Health Research Institute, University of Alberta, Edmonton, Canada).

Suspension or premature termination of the clinical investigation The sponsor/principal investigator and the ethics committees can make decisions about trial discontinuation. If the trial is terminated or suspended the parents of all trial participants will be informed and appropriate follow-up will be assured. If sponsor/principal investigator terminates or suspends the trial the relevant ethics committees will be provided with a detailed written explanation of the termination or suspension.

The sponsor/principal investigator can, upon completion of the analysis of the reason(s) for a suspension, decide to lift the suspension when the necessary corrective actions have been implemented. The investigators and ethics committees will be notified and provided with the relevant data supporting the decision.

Stopping rules

The DSMB will review the data at interim analyses at 10%, 25% and 50%. Predefined stopping rules will include:

1. An increased mortality in the SI+CC group by 25% compared to the 3:1 C:V group at the predefined interim analysis at 10%, 25% and 50%.
2. Increase in rate of morbidities including pneumothorax, intraventricular hemorrhage or the combination, in the SI+CC group by 25% compared to the 3:1 C:V group at the predefined interim analysis at 10%, 25% and 50%.
3. Bayesian posterior probability of SI+CC group being better than the control is less than 0.5 or greater than 0.98. (Posterior probability of SI+CC arm to reduce time to ROSC by 10% or more compared to the control arm will be calculated. If this probability is less than 0.5, the trial will be stopped for futility. If the posterior probability is greater than 0.98, DSMB will consider the trial to be stopped for superiority. Since no statistical tests will be performed at interim analyses, type I error (alpha) does not need adjustment).

Opt-out Rule In any cases were CPR is ongoing for 5 minutes, the clinical team must convert to the standard method of care using the 3:1 C:V ratio.

Ethical Considerations The SURV1VE-trial will be conducted in compliance with the guidelines of the Declaration of Helsinki in its latest form, the International Conference on Harmonization of Good Clinical Practice Guidelines. In case of modifications in the study protocol that are not merely of a formal nature but contain changes pertinent to the study participants, a renewed vote of the relevant ethics committees will be obtained. If applicable, the patients (parents) will be informed in the patient information and consent form about changes in the terms and conditions of the trial. The SURV1VE-trial will only start the randomization of participants after approvals from the relevant ethics committees have been obtained.

Data management Data handling and archiving Source data will be registered in the participant's medical records/CRF and into the eCRF. A common web-based eCRF will be devised to enable a central database (Women and Children's Health Research Institute, University of Alberta, Edmonton, Canada). Data entry into the central database and handling of medical records is the responsibility of the investigators. After the establishment of a 'clean file', the database will be locked; The data will be locked after completion of patient recruitment and data entry. After long-term follow-up data entry this portion of the database will locked. Data will be stored for statistical analysis at the Biostatistics Unit, Women and Children's Health Research Institute, University of Alberta, Edmonton, Canada. The trial database will hereafter be kept according to the respective national laws. After the end of trial, the data will be archived for 25 years according to good clinical practice guidelines. At each trial-site the data flow will be monitored according to the GCP principles by a locally appointed external monitoring committee. After completion of statistical data analysis, data will be pseudo-anonymized and stored at the University of Alberta, Edmonton, Canada.

Data protection The investigator(s) permits trial-related monitoring, audits, and regulatory inspection(s) by providing direct access to the source data and other relevant documents. Trial data will be handled according to regulations of the data protection agency in the respective countries.

Quality assurance The trial will be carried out in accordance with the Declaration of Helsinki in its latest form and the International Conference on Harmonization Good Clinical Practice (ICH-GCP) guidelines.

Monitoring The chief investigator consents to data evaluation being performed by the person in charge of monitoring in accordance with the monitoring plan, in order to ensure satisfactory data collection and adherence to the study protocol. Furthermore, the chief investigator states that he/she is willing to cooperate with this person and shall provide this person with all required information whenever necessary. This includes access to all documents related to the trial, including study-relevant medical files of patients in original form. The tasks of the investigator include maintenance of these patients' medical files as comprehensively as possible; this includes information concerning medical history, accompanying diseases, inclusion in the trial, data about visits, results of investigations, dispensing of medication, and adverse events. The monitor will also be permitted to perform data evaluation and draw comparisons with the relevant medical files in accordance with the standard operating procedures and ICH-GCP guidelines at predetermined intervals, in order to ensure adherence to the study protocol and continuous registration of data. All original medical reports required as sources for the information given in the CRF or the database shall be inspected. The study participants will have given their consent to such inspection by signing the consent form. The person in charge of monitoring is obliged to treat all information as confidential and to preserve the basic claims of the study participants in respect of integrity and protection of their privacy.

ELIGIBILITY:
Inclusion Criteria:

* Infants (term or preterm infants >28 weeks' gestation) requiring CC in the delivery room will be eligible for the trial.

Exclusion Criteria:

* Infants will be excluded if they have a congenital abnormality or condition that might have an adverse effect on breathing or ventilation (e.g. congenital diaphragmatic hernia), or congenital heart disease requiring intervention in the neonatal period. Infants would be also excluded if their parents refused to give consent to this study.

Ages: 0 Minutes to 20 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schmolzer, Principal Investigator — University of Alberta
Locations (4):
- Austria (2):
  - Medical University Graz, Graz
  - Medical University Vienna, Vienna
- Canada (2):
  - Royal Alexandra Hospital, Edmonton
  - IWK Health Centre, Halifax

REFERENCES:
- [Background] Perlman JM, Wyllie J, Kattwinkel J, Wyckoff MH, Aziz K, Guinsburg R, Kim HS, Liley HG, Mildenhall L, Simon WM, Szyld E, Tamura M, Velaphi S; Neonatal Resuscitation Chapter Collaborators. Part 7: Neonatal Resuscitation: 2015 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Circulation. 2015 Oct 20;132(16 Suppl 1):S204-41. doi: 10.1161/CIR.0000000000000276. No abstract available. PMID 26472855
- [Background] Wyckoff MH, Aziz K, Escobedo MB, Kapadia VS, Kattwinkel J, Perlman JM, Simon WM, Weiner GM, Zaichkin JG. Part 13: Neonatal Resuscitation: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S543-60. doi: 10.1161/CIR.0000000000000267. No abstract available. PMID 26473001
- [Background] Wyllie J, Perlman JM, Kattwinkel J, Wyckoff MH, Aziz K, Guinsburg R, Kim HS, Liley HG, Mildenhall L, Simon WM, Szyld E, Tamura M, Velaphi S; Neonatal Resuscitation Chapter Collaborators. Part 7: Neonatal resuscitation: 2015 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science with Treatment Recommendations. Resuscitation. 2015 Oct;95:e169-201. doi: 10.1016/j.resuscitation.2015.07.045. Epub 2015 Oct 15. No abstract available. PMID 26477424
- [Background] Schmolzer GM, O Reilly M, Fray C, van Os S, Cheung PY. Chest compression during sustained inflation versus 3:1 chest compression:ventilation ratio during neonatal cardiopulmonary resuscitation: a randomised feasibility trial. Arch Dis Child Fetal Neonatal Ed. 2018 Sep;103(5):F455-F460. doi: 10.1136/archdischild-2017-313037. Epub 2017 Oct 7. PMID 28988159
- [Background] Li ES, Gorens I, Cheung PY, Lee TF, Lu M, O'Reilly M, Schmolzer GM. Chest Compressions during Sustained Inflations Improve Recovery When Compared to a 3:1 Compression:Ventilation Ratio during Cardiopulmonary Resuscitation in a Neonatal Porcine Model of Asphyxia. Neonatology. 2017;112(4):337-346. doi: 10.1159/000477998. Epub 2017 Aug 3. PMID 28768280
- [Background] Solevag AL, Schmolzer GM. Optimal Chest Compression Rate and Compression to Ventilation Ratio in Delivery Room Resuscitation: Evidence from Newborn Piglets and Neonatal Manikins. Front Pediatr. 2017 Jan 23;5:3. doi: 10.3389/fped.2017.00003. eCollection 2017. PMID 28168185
- [Background] Li ES, Cheung PY, Lee TF, Lu M, O'Reilly M, Schmolzer GM. Return of spontaneous Circulation Is Not Affected by Different Chest Compression Rates Superimposed with Sustained Inflations during Cardiopulmonary Resuscitation in Newborn Piglets. PLoS One. 2016 Jun 15;11(6):e0157249. doi: 10.1371/journal.pone.0157249. eCollection 2016. PMID 27304210
- [Background] Sobotka KS, Hooper SB, Crossley KJ, Ong T, Schmolzer GM, Barton SK, McDougall AR, Miller SL, Tolcos M, Klingenberg C, Polglase GR. Single Sustained Inflation followed by Ventilation Leads to Rapid Cardiorespiratory Recovery but Causes Cerebral Vascular Leakage in Asphyxiated Near-Term Lambs. PLoS One. 2016 Jan 14;11(1):e0146574. doi: 10.1371/journal.pone.0146574. eCollection 2016. PMID 26765258
- [Background] Solevag AL, Cheung PY, O'Reilly M, Schmolzer GM. A review of approaches to optimise chest compressions in the resuscitation of asphyxiated newborns. Arch Dis Child Fetal Neonatal Ed. 2016 May;101(3):F272-6. doi: 10.1136/archdischild-2015-309761. Epub 2015 Dec 1. PMID 26627554
- [Background] Solevag AL, Cheung PY, Lie H, O'Reilly M, Aziz K, Nakstad B, Schmolzer GM. Chest compressions in newborn animal models: A review. Resuscitation. 2015 Nov;96:151-5. doi: 10.1016/j.resuscitation.2015.08.001. Epub 2015 Aug 19. PMID 26296585
- [Background] Li ES, Cheung PY, O'Reilly M, Schmolzer GM. Change in tidal volume during cardiopulmonary resuscitation in newborn piglets. Arch Dis Child Fetal Neonatal Ed. 2015 Nov;100(6):F530-3. doi: 10.1136/archdischild-2015-308363. Epub 2015 Jul 1. PMID 26139543
- [Background] Sobotka KS, Polglase GR, Schmolzer GM, Davis PG, Klingenberg C, Hooper SB. Effects of chest compressions on cardiovascular and cerebral hemodynamics in asphyxiated near-term lambs. Pediatr Res. 2015 Oct;78(4):395-400. doi: 10.1038/pr.2015.117. Epub 2015 Jun 18. PMID 26086644
- [Background] Schmolzer GM, Kumar M, Aziz K, Pichler G, O'Reilly M, Lista G, Cheung PY. Sustained inflation versus positive pressure ventilation at birth: a systematic review and meta-analysis. Arch Dis Child Fetal Neonatal Ed. 2015 Jul;100(4):F361-8. doi: 10.1136/archdischild-2014-306836. Epub 2014 Dec 30. PMID 25550472
- [Background] Li ES, Cheung PY, Pichler G, Aziz K, Schmolzer GM. Respiratory function and near infrared spectroscopy recording during cardiopulmonary resuscitation in an extremely preterm newborn. Neonatology. 2014;105(3):200-4. doi: 10.1159/000357609. Epub 2014 Jan 24. PMID 24481290
- [Background] Schmolzer GM, O'Reilly M, Labossiere J, Lee TF, Cowan S, Nicoll J, Bigam DL, Cheung PY. 3:1 compression to ventilation ratio versus continuous chest compression with asynchronous ventilation in a porcine model of neonatal resuscitation. Resuscitation. 2014 Feb;85(2):270-5. doi: 10.1016/j.resuscitation.2013.10.011. Epub 2013 Oct 22. PMID 24161768
- [Background] Schmolzer GM, O'Reilly M, Labossiere J, Lee TF, Cowan S, Qin S, Bigam DL, Cheung PY. Cardiopulmonary resuscitation with chest compressions during sustained inflations: a new technique of neonatal resuscitation that improves recovery and survival in a neonatal porcine model. Circulation. 2013 Dec 3;128(23):2495-503. doi: 10.1161/CIRCULATIONAHA.113.002289. Epub 2013 Oct 2. PMID 24088527
- [Background] Solevag AL, Lee TF, Lu M, Schmolzer GM, Cheung PY. Tidal volume delivery during continuous chest compressions and sustained inflation. Arch Dis Child Fetal Neonatal Ed. 2017 Jan;102(1):F85-F87. doi: 10.1136/archdischild-2016-311043. Epub 2016 Aug 26. PMID 27566670
- [Background] Boldingh AM, Solevag AL, Aasen E, Nakstad B. Resuscitators who compared four simulated infant cardiopulmonary resuscitation methods favoured the three-to-one compression-to-ventilation ratio. Acta Paediatr. 2016 Aug;105(8):910-6. doi: 10.1111/apa.13339. Epub 2016 Feb 18. PMID 26801948
- [Background] Dannevig I, Solevag AL, Saugstad OD, Nakstad B. Lung Injury in Asphyxiated Newborn Pigs Resuscitated from Cardiac Arrest - The Impact of Supplementary Oxygen, Longer Ventilation Intervals and Chest Compressions at Different Compression-to-Ventilation Ratios. Open Respir Med J. 2012;6:89-96. doi: 10.2174/1874306401206010089. Epub 2012 Sep 20. PMID 23115599
- [Background] Solevag AL, Madland JM, Gjaerum E, Nakstad B. Minute ventilation at different compression to ventilation ratios, different ventilation rates, and continuous chest compressions with asynchronous ventilation in a newborn manikin. Scand J Trauma Resusc Emerg Med. 2012 Oct 17;20:73. doi: 10.1186/1757-7241-20-73. PMID 23075128
- [Background] Solevag AL, Dannevig I, Wyckoff M, Saugstad OD, Nakstad B. Return of spontaneous circulation with a compression:ventilation ratio of 15:2 versus 3:1 in newborn pigs with cardiac arrest due to asphyxia. Arch Dis Child Fetal Neonatal Ed. 2011 Nov;96(6):F417-21. doi: 10.1136/adc.2010.200386. Epub 2011 Mar 10. PMID 21393311
- [Background] Dannevig I, Solevag AL, Wyckoff M, Saugstad OD, Nakstad B. Delayed onset of cardiac compressions in cardiopulmonary resuscitation of newborn pigs with asphyctic cardiac arrest. Neonatology. 2011;99(2):153-62. doi: 10.1159/000302718. Epub 2010 Sep 11. PMID 20829634
- [Background] Solevag AL, Dannevig I, Wyckoff M, Saugstad OD, Nakstad B. Extended series of cardiac compressions during CPR in a swine model of perinatal asphyxia. Resuscitation. 2010 Nov;81(11):1571-6. doi: 10.1016/j.resuscitation.2010.06.007. Epub 2010 Jul 17. PMID 20638769
- [Background] Chandra N, Rudikoff M, Weisfeldt ML. Simultaneous chest compression and ventilation at high airway pressure during cardiopulmonary resuscitation. Lancet. 1980 Jan 26;1(8161):175-8. doi: 10.1016/s0140-6736(80)90662-5. PMID 6101633
- [Background] Tsui BC, Horne S, Tsui J, Corry GN. Generation of tidal volume via gentle chest pressure in children over one year old. Resuscitation. 2015 Jul;92:148-53. doi: 10.1016/j.resuscitation.2015.02.021. Epub 2015 Mar 4. PMID 25749553
- [Background] Babbs CF, Meyer A, Nadkarni V. Neonatal CPR: room at the top--a mathematical study of optimal chest compression frequency versus body size. Resuscitation. 2009 Nov;80(11):1280-4. doi: 10.1016/j.resuscitation.2009.07.014. Epub 2009 Aug 27. PMID 19713026
- [Background] Hemway RJ, Christman C, Perlman J. The 3:1 is superior to a 15:2 ratio in a newborn manikin model in terms of quality of chest compressions and number of ventilations. Arch Dis Child Fetal Neonatal Ed. 2013 Jan;98(1):F42-5. doi: 10.1136/archdischild-2011-301334. Epub 2012 Apr 3. PMID 22491015
- [Background] Srikantan SK, Berg RA, Cox T, Tice L, Nadkarni VM. Effect of one-rescuer compression/ventilation ratios on cardiopulmonary resuscitation in infant, pediatric, and adult manikins. Pediatr Crit Care Med. 2005 May;6(3):293-7. doi: 10.1097/01.PCC.0000161621.74554.15. PMID 15857527
- [Background] Kern KB, Hilwig RW, Berg RA, Sanders AB, Ewy GA. Importance of continuous chest compressions during cardiopulmonary resuscitation: improved outcome during a simulated single lay-rescuer scenario. Circulation. 2002 Feb 5;105(5):645-9. doi: 10.1161/hc0502.102963. PMID 11827933
- [Derived] Schmolzer GM, Pichler G, Solevag AL, Law BHY, Mitra S, Wagner M, Pfurtscheller D, Yaskina M, Cheung PY; SURV1VE- Trial Investigators. Sustained inflation and chest compression versus 3:1 chest compression to ventilation ratio during cardiopulmonary resuscitation of asphyxiated newborns (SURV1VE): A cluster randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2024 Jun 19;109(4):428-435. doi: 10.1136/archdischild-2023-326383. PMID 38212104
- [Derived] Schmolzer GM, Pichler G, Solevag AL, Fray C, van Os S, Cheung PY; SURV1VE trial collaborators. The SURV1VE trial-sustained inflation and chest compression versus 3:1 chest compression-to-ventilation ratio during cardiopulmonary resuscitation of asphyxiated newborns: study protocol for a cluster randomized controlled trial. Trials. 2019 Feb 19;20(1):139. doi: 10.1186/s13063-019-3240-8. PMID 30782199

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention (CC+SI): Infants randomized into the "CC+SI group" will receive a SI with a PIP of 25-30 cmH2O while receiving chest compression. The SI will be delivered over a period of 45 seconds. This will be followed by PEEP of 5-8 cm water to perform an assessment of the newborn's heart rate. If heart rate is >60/min continue with standard care as per local hospital policy (standard hospital practice guideline). If heart rate remains <60/min continue with CC+SI for another 45sec at which time a further assessment should be performed. If heart rate remains <60/min continue with CC+SI.
  CC+SI: chest compression will be delivered during sustained inflation (CC+SI). The duration of each sustain inflation is 20sec. After 20sec a pause of 1sec id done before the next sustained inflation is delivered for another 20sec. Chest compressions are given continuously. This approach is continued for a max of 5 minutes, when the team has to switch to 3:1 C:V.
Period: Overall Study
Arm/Group | Intervention (CC+SI) | Control (3:1 C:V)
Started | 12 | 15
Completed | 11 | 14
Not Completed | 1 | 1
Not completed — Declined consent | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention (CC+SI) | Control (3:1 C:V) | Total
Number analyzed (Participants) | 11 | 14 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 14 | 25
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 7 | 7 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Return of Spontaneous Circulation
Description: Duration of chest compression heart rate is >60/min for 60sec.
Time Frame: up to 60 Minutes of chest compression
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Intervention (CC+SI) | Control (3:1 C:V)
Number analyzed (Participants) | 11 | 14
seconds | 90 [60 to 270] | 615 [174 to 780]

2. Secondary Outcome: Mortality
Description: Number of infants who die until discharge - comparison between group
Time Frame: Until infant is discharge from hospital (maximum of 30 weeks after birth)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (CC+SI) | Control (3:1 C:V)
Number analyzed (Participants) | 11 | 14
Participants | 2 | 8

3. Secondary Outcome: Rate of Brain Injury - Intraventricular Hemorrhage
Description: Brain injury either by ultrasound or magnet resonance imaging - comparison between group
Time Frame: Until infant is discharge from hospital (maximum of 30 weeks after birth)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (CC+SI) | Control (3:1 C:V)
Number analyzed (Participants) | 11 | 14
Participants | 1 | 2

4. Secondary Outcome: Necrotizing Enterocolitis
Description: Number of infants who develop Necrotizing enterocolitis - comparison between group
Time Frame: Until infant is discharge from hospital (maximum of 30 weeks after birth)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (CC+SI) | Control (3:1 C:V)
Number analyzed (Participants) | 11 | 14
Participants | 0 | 0

5. Secondary Outcome: Epinephrine Doses Via Umbilical Venous Catheter
Description: Epinephrine Doses via Umbilical venous catheter
Time Frame: during resuscitation at birth
Measure: Mean (Standard Deviation); unit: Doses
Arm/Group | Intervention (CC+SI) | Control (3:1 C:V)
Number analyzed (Participants) | 11 | 14
Doses | 2.3 (1.5) | 2 (1.4)

ADVERSE EVENTS:
Time Frame: Until infant is discharge from hospital (maximum of 30 weeks after birth)
Arm/Group | Intervention (CC+SI) | Control (3:1 C:V)
All-Cause Mortality (participants affected / at risk) | 2/11 | 8/14
Serious Adverse Events (participants affected / at risk) | 2/11 | 4/14
Other Adverse Events (participants affected / at risk) | 0/11 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (CC+SI) (N=11) | Control (3:1 C:V) (N=14)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
intraventricular hemorrhage (Nervous system disorders) | 1 (1) | 2 (2) — intraventricular hemorrhage garde 3 and 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT02858583/Prot_SAP_000.pdf